CLINICAL TRIAL: NCT01829425
Title: Protocol for Brain-Centered Therapy Versus Medication for Urgency Urinary Incontinence An RCT: Hypnotherapy Or Pharmacotherapy
Brief Title: Brain-Centered Therapy Versus Medication for Urgency Urinary Incontinence : Hypnotherapy Or Pharmacotherapy
Acronym: Hyp-hOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Yuko Komesu, MD, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-314; 1R01AT007171-01A1 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Urinary Incontinence, Urge
Keywords: Hypnosis; Mind-Body Therapy; Anticholinergics; Female Urogenital Diseases
MeSH Terms: conditions — Urinary Incontinence, Urge; Female Urogenital Diseases | interventions — Tolterodine Tartrate; oxybutynin; Hypnosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anticholinergic medications (Active Comparator): Either of two standard, long acting anti-cholinergic medications (Long acting Tolterodine or Extended Release Oxybutynin)will be given. Subjects receive 8 weeks of medication counseling in conjunction with the medications. Medications will be continued for 1 year.
  Interventions: Drug: Anticholinergic medications
- Hypnotherapy (Active Comparator): Subjects will receive approximately weekly hypnotherapy sessions over 8 weeks and will receive/download digital recordings for home practice. Subjects will be encouraged to practice self-hypnosis +/or listen to their recordings for 1 year.
  Interventions: Behavioral: Hypnotherapy

INTERVENTIONS:
Drug: Anticholinergic medications — The study will use either of two standard, long acting anti-cholinergic medications and dosages. Pharmacotherapy counseling sessions will also be administered over 8 weeks by trained research personnel. Pharmacotherapy counseling sessions will be audio-recorded and one or more sessions will be reviewed by study personnel to ensure that the medication counselor administers the sessions in a standardized fashion. Pill counts will be performed at the conclusion of the 8 weeks of pharmacotherapy counseling. Subjects will be provided the medication for 1 year.
  Other Names: Tolterodine (Detrol LA or equivalent generic); Oxybutynin (Ditropan Extended Release or equivalent generic)
  Arms: Anticholinergic medications
Behavioral: Hypnotherapy — Hypnotherapy will be administered approximately weekly over 8 weeks by certified, trained clinical hypnotherapists. Sessions will be audio-recorded and one or more sessions will be reviewed by study personnel to ensure that the hypnotherapist administers the hypnotherapy session in a standardized fashion.Subjects will receive or download a digital recording specially prepared for them to for home practice of hypnotherapy sessions.Following the 8 weeks of therapy, subjects will be encouraged to continue to practice self-hypnosis and/or listen to their home practice digital recording and this practice will be tracked for the 1 year duration of the study.
  Arms: Hypnotherapy

SUMMARY:
This study is randomized controlled trial in which urgency incontinent women (approximately 150-160) will be randomized to hypnotherapy or pharmacotherapy and evaluated at months 2, 6 &12 Hypotheses: Among patients with urgency urinary incontinence (UUI), hypnotherapy will be non-inferior pharmacotherapy in diminishing UUI episodes. Hypnotherapy may be superior or may not differ from pharmacotherapy in diminishing symptoms or quality of life based on validated questionnaires and/or other diary parameters.

DETAILED DESCRIPTION:
Study Objectives Primary: To compare change in Urgency Urinary Incontinence (UUI) episodes at 2 month follow-up on voiding diaries between hypnotherapy and pharmacotherapy groups (to determine whether hypnotherapy is at least as effective and durable in treating UUI as pharmacotherapy)

Secondary Analyses:

* To determine whether hypnotherapy is at least as effective in treating UUI as pharmacotherapy comparing change in UUI episodes on voiding diary at 6 and 12 month follow-up
* To determine whether hypnotherapy differs from pharmacotherapy in treating UUI comparing change in questionnaire results and urinary frequency
* enrolled following administration of the Overactive Bladder (OAB) Awareness tool. Participants will keep voiding diaries then be randomized to either pharmacotherapy and conventional behavioral therapy or hypnotherapy and conventional behavioral therapy. Approximately 150-160 women will be randomized.

Randomization will occur using a computer-generated randomization scheme in varying permuted block sizes. Study personnel performing data entry will be masked to participants' treatment. Masking participants to treatment is not feasible. Participants will be followed at 2,6 & 12 months. Measurements will be performed before treatment, following completion of treatment visits (approximately 8 weeks), and at 6 and 12 months. Primary analysis will be intention to treat. Exploratory analyses of secondary outcomes will also be performed.

Study Visits: UUI participant screening: Study information given. Screening questionnaire given. Visit 1 Enrollment: Formal screening for eligibility, voiding diary reviewed, if eligible, written consent obtained with administration of study questionnaires, demographic and past medical history administration forms, Pelvic Organ Prolapse Quantitation (POP-Q) exam & hypnotic susceptibility testing scheduled. Pariticipants undergo hypnotic susceptibility testing prior to randomization. Participants randomized to treatment and contacted, treatments arranged. Hypnotherapy group: undergo weekly treatments over 8 weeks. Pharmacotherapy group: weekly counseling sessions over 8 week: Following hypnotherapy or medication counseling completion, f/u voiding diaries collected & study questionnaires administered. One of two long acting anti-cholinergic medications offered (Long acting Tolterodine or Extended Release Oxybutynin or equivalent generic substitutes).

6 & 12 month follow-up: Pharmacotherapy subjects receive medications for 1 year and Hypnotherapy subjects encouraged to continue self-hypnosis for 1 year with assistance of audio-recordings, with 1 optional hypnotherapy session between 6-12 months..

Participants informed pharmacotherapy & hypnotherapy sessions are audio-recorded and reviewed ensuring manual of procedures are followed.

ELIGIBILITY:
Inclusion Criteria:(For randomized trial)

1. Non-pregnant English-speaking women
2. 18 yo or older
3. Overactive Bladder (OAB) Awareness scores ≥ 8
4. 3 UUI episodes/week for ≥ 3 months

Exclusion Criteria: (For Randomized trial)

1. Women with a history of neurologic diseases such as Multiple Sclerosis, Parkinson's disease, stroke, or dementia
2. History of schizophrenia or untreated bipolar disorder or current drug or alcohol dependence
3. Women who have taken anticholinergic medications for UUI within the last 3 weeks (women who have taken anti-cholinergics for UUI but discontinued them > than 3 weeks ago may participate in the study) or have a sacral neuromodulator in place to treat UUI or have received Onabotulinum toxin A in the last 12 months to treat UUI
4. Contraindications to anticholinergic medications (untreated narrow angle glaucoma, significant urinary retention or gastric retention)
5. Pregnant women or lactating women, women who plan to become pregnant in the next year, or pre-menopausal women unwilling to use contraception if engaging in sexual relations during the year of study participation (hysterectomy is considered to be a form of contraception)
6. Untreated urinary tract infection
7. Prolapse which extends past the hymen (POP-Q points of ≥ 1+) which may be responsible for UUI symptoms
8. Women who cannot keep the majority of the study therapy appointments or those without reliable contact phone numbers or methods of communication with the study personnel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Komesu, MD, Principal Investigator — University of New Mexcio Health Science Center
Locations (1):
- University of New Mexico Health Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
The information will be shared with other researchers upon their request. Our IRB required that we re-consent participants in order to make their data available to others. We can only share the information available on participants who signed these additional consents.
Supporting Information: Study Protocol
Time Frame: 6 months after manuscript for the primary outcome is accepted for publication. Anticipated time for manuscript acceptance July 2019. Anticipated availability 3-5 years.
Access Criteria: Dr. Komesu and Dr. Ketai will review requests. Access criteria includes de-identified dataset (including de-identification of dates of visit as this may be interpreted as a potential identifier) of those who consented to have data shared. Data for secondary manuscripts in progress by PIs will be shared only after PIs publish said data 6 months post-publication.

REFERENCES:
- [Background] Komesu YM, Ketai LH, Mayer AR, Teshiba TM, Rogers RG. Functional MRI of the Brain in Women with Overactive Bladder: Brain Activation During Urinary Urgency. Female Pelvic Med Reconstr Surg. 2011;17(1):50-54. doi: 10.1097/SPV.0b013e3182065507. PMID 21399722
- [Background] Komesu YM, Sapien RE, Rogers RG, Ketai LH. Hypnotherapy for treatment of overactive bladder: a randomized controlled trial pilot study. Female Pelvic Med Reconstr Surg. 2011 Nov;17(6):308-13. doi: 10.1097/SPV.0b013e31823a08d9. PMID 22453228
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Sandvik H, Seim A, Vanvik A, Hunskaar S. A severity index for epidemiological surveys of female urinary incontinence: comparison with 48-hour pad-weighing tests. Neurourol Urodyn. 2000;19(2):137-45. doi: 10.1002/(sici)1520-6777(2000)19:23.0.co;2-g. PMID 10679830
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] Coyne KS, Zyczynski T, Margolis MK, Elinoff V, Roberts RG. Validation of an overactive bladder awareness tool for use in primary care settings. Adv Ther. 2005 Jul-Aug;22(4):381-94. doi: 10.1007/BF02850085. PMID 16418145
- [Background] Burgio KL, Locher JL, Goode PS, Hardin JM, McDowell BJ, Dombrowski M, Candib D. Behavioral vs drug treatment for urge urinary incontinence in older women: a randomized controlled trial. JAMA. 1998 Dec 16;280(23):1995-2000. doi: 10.1001/jama.280.23.1995. PMID 9863850
- [Derived] Ketai LH, Komesu YM, Schrader RM, Rogers RG, Sapien RE, Dodd AB, Mayer AR. Mind-body (hypnotherapy) treatment of women with urgency urinary incontinence: changes in brain attentional networks. Am J Obstet Gynecol. 2021 May;224(5):498.e1-498.e10. doi: 10.1016/j.ajog.2020.10.041. Epub 2020 Oct 26. PMID 33122028
- [Derived] Komesu YM, Schrader RM, Rogers RG, Sapien RE, Mayer AR, Ketai LH. Hypnotherapy or medications: a randomized noninferiority trial in urgency urinary incontinent women. Am J Obstet Gynecol. 2020 Feb;222(2):159.e1-159.e16. doi: 10.1016/j.ajog.2019.08.025. Epub 2019 Aug 23. PMID 31449805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited March 2013 through October 2016 from the UNMH Urogynecology clinics
Pre-assignment Details: Patients required to keep 3 day voiding diary to confirm their eligibility for the study prior to randomization. Pts also underwent hypnotic susceptibility testing prior to randomization.
  Of those consented, 13 did not go on to randomization: 8 were excluded because they did not meet inclusion criteria and 5 were lost to further followup
Period: Overall Study
Arm/Group | Anticholinergic Medications | Hypnotherapy
Started | 78 | 74
Completed | 72 (completed primary outcome 2 month f/u N=72) | 70 (completed primary outcome 2 month f/u N=70)
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: analysis was performed on baseline of patients with primary outcome data; baseline analysis includes the 70 and 72 patients with 2 month data
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypnotherapy | Anticholinergic Medications | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.77) | 59.5 (10.30) | 58.55 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 142
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 15 | 39
  Not Hispanic or Latino | 45 | 55 | 100
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 52 | 61 | 113
  More than one race | 11 | 7 | 18
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 70 | 72 | 142
Urgency Incontinence episodes on 3 day diary [Median (Inter-Quartile Range); unit: episodes] | 8 [4 to 14] | 7 [4 to 11] | 7.5 [4 to 13]
Overactive bladder short form (OABq-SF) questionnaires [Mean (Standard Deviation); unit: units on a scale] — Lower scores on the bother sub-scale are better (less bother) and Higher scores on the quality of life sub-scale are better (higher quality of life) ; validated questionnaire scores for both Sub-scales range from 0-100. These results are stand-alone; they are not combined
  units on a scale
    Overactive Bladder Questionnaire Short Form Bother | 66.88 (21.26) | 66.99 (21.60) | 66.94 (21.43)
    Overactive Bladder Short Form Quality of Life | 47.11 (27.40) | 50.38 (25.29) | 48.75 (26.35)
number of voids on bladder diary [Mean (Standard Deviation); unit: episodes] — Patients recorded their number of voids (total) on a 3-day bladder diary
  episodes | 29.07 (8.71) | 29.19 (8.43) | 29.13 (8.57)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Urgency Urinary Incontinence Episodes
Description: Percent change in UUI episodes from baseline to 2 months with comparison made between hypnotherapy & pharmacotherapy
Time Frame: Baseline and 2 month follow-up
Population: Randomized patients with primary outcome (diary information) 2 months. Hypnotherapy: 74 randomized; of those randomized 3 had withdrawn, 1 was lost=70 with primary outcome information for analysis. Medications: 78 randomized-- 4 withdrawn. 2 were missing diary information=72 with primary outcome information for analysis
Measure: Median (95% Confidence Interval); unit: percentage change in median UUI episodes
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 70 | 72
percentage change in median UUI episodes | 73 [60 to 88.9] | 88.6 [78.6 to 100]
Statistical Analysis 1: Comparison: Hypnotherapy vs Anticholinergic Medications; Test type: Non-Inferiority — The study design will use a non-inferiority design to compare the primary outcome (change in UUI episodes in the hypnotherapy versus pharmacotherapy groups). With respect to the outcome variable of percent reduction in UUI episodes as determined by bladder diaries, we will use a one-sided non- inferiority test at level alpha = 0.25 and a non-inferiority margin of 5%; p < .025, Exact Mann Whitney; Due dispersion, medians were calculated. Exact Mann Whitney test was used for this analysis; Difference in median % change between gr = 5, 95% CI 1-sided [lower limit 5] — Hypnotherapy - Pharmacotherapy. % difference in median % change in UUI episodes with lower bounds > - 5% would be consistent with non-inferiority

2. Secondary Outcome: Percent Change in Urgency Urinary Incontinence Episodes
Description: Differences comparing hypnotherapy to pharmacotherapy percent change in median UUI episodes
Time Frame: 6 months
Population: At 6 months. Hypnotherapy: 74 women randomized-- 4 withdrawn, 2 lost and 1 missing diary information=67 analyzed with diary data. Medication: 78 randomized, 6 had withdrawn and 1 lost=71 analyzed with diary data
Measure: Median (95% Confidence Interval); unit: percentage change in median UUI episodes
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 67 | 71
percentage change in median UUI episodes | 85.7 [75 to 100] | 83.3 [64.7 to 100]
Statistical Analysis 1: Comparison: Hypnotherapy vs Anticholinergic Medications; Test type: Non-Inferiority — The study design will use a non-inferiority design to compare the primary outcome (change in UUI episodes in the hypnotherapy versus pharmacotherapy groups). With respect to the outcome variable of percent reduction in UUI episodes as determined by bladder diaries, we will use a one-sided non- inferiority test at level alpha = 0.25 and a non-inferiority margin of 5%. If; p < .025, Exact Mann Whitney; Difference in median % change between gr = 5, 95% CI 1-sided [lower limit 5]

3. Secondary Outcome: Percent Change in Urgency Urinary Incontinence Episodes
Description: Percent change in median UUI episodes from baseline to 12 months with comparison made between hypnotherapy & pharmacotherapy
Time Frame: 12 months
Population: Pts with diary data at 12 months. For the Hypnotherapy group, of the 74 women randomized, 4 had withdrawn and 1 was missing diary data. For the medication group, of the 78 women randomized, 7 had withdrawn.
Measure: Median (95% Confidence Interval); unit: percentage change in median UUI episodes
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 69 | 71
percentage change in median UUI episodes | 85.7 [66.7 to 94.4] | 80.0 [54.5 to 100.0]

4. Secondary Outcome: Overactive Bladder Questionnaire Short Form Symptom Bother
Description: Overactive Bladder Questionnaire Short Form symptom bother Scale. Sub-Scale range 0-100. Higher numbers are worse (more bother) and lower numbers are better (less bother)
Time Frame: 2 months
Population: Randomized patients with primary outcome (diary information) 2 months. Hypnotherapy: 70 had diary information; of those randomized 3 had withdrawn, 1 was lost=70 with primary outcome information for analysis. Medications: 78 randomized-- 4 withdrawn. 2 were missing diary information=72 with primary outcome information for analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a sub-scale
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 70 | 72
scores on a sub-scale | 38.17 [30.19 to 46.14] | 35.33 [28.64 to 42.02]

5. Secondary Outcome: Overactive Bladder Questionnaire Short Form Symptom Bother
Description: Overactive Bladder Questionnaire Short Form symptom bother. Sub-scale range 0-100. Higher numbers are worse (more bother) and lower numbers are better (less bother)
Time Frame: 6 months
Population: At 6 months in the hypnotherapy group, 4 had withdrawn and 2 were lost and 1 missing diary. In the medication group, 6 had withdrawn and 1 was missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: sub-scale scores
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 67 | 71
sub-scale scores | 34.61 [26.26 to 42.96] | 27.93 [20.66 to 35.20]

6. Secondary Outcome: Overactive Bladder Questionnaire Short Form Symptom Bother
Description: as for outcome 5
Time Frame: 12 months
Population: 12 months. Hypnotherapy: 74 randomized, 4 withdrawn & 1 was missing diary=69 analyzed with diary data. Medication: 78 randomized, 7 had withdrawn=71 analyzed with diary data.
Measure: Least Squares Mean (95% Confidence Interval); unit: sub-scale scores
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 69 | 71
sub-scale scores | 32.27 [22.89 to 41.66] | 30.74 [22.53 to 38.95]

7. Secondary Outcome: Overactive Bladder Questionnaire Short Form Quality of Life
Description: Overactive Bladder questionnaire-Short Form Quality of Life. Higher scores are better (better quality of life) and lower scores are worse (poorer quality of life). sub-score range 0-100.
Time Frame: 2 months
Population: Randomized patients with primary outcome (diary information) 2 months. Hypnotherapy: 74 randomized; 3 withdrawn, 1 lost=70 with primary outcome information used for analysis for secondary outcomes. Medications: 78 randomized-- 4 withdrawn, 2 were missing diary information=72 for analysis of secondary outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: sub-scale scores
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 70 | 72
sub-scale scores | 73.96 [66.93 to 81.00] | 74.86 [68.96 to 80.76]

8. Secondary Outcome: Overactive Bladder Questionnaire Short Form Quality of Life
Description: Overactive Bladder questionnaire Short Form Quality of Life. Higher scores are better (better quality of life) and lower scores are worse (poorer quality of life). sub-scale score range 0-100.
Time Frame: 6 months
Population: At 6 months, in the hypnotherapy group: 4 had withdrawn and 2 were lost and 1 missing diary. In the medication group: 6 had withdrawn and 1 was lost.
Measure: Least Squares Mean (95% Confidence Interval); unit: sub-scale scores
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 67 | 71
sub-scale scores | 75.85 [68.24 to 83.46] | 80.19 [73.63 to 86.75]

9. Secondary Outcome: Overactive Bladder Questionnaire Short Form Quality of Life
Description: Overactive Bladder questionnaire-Short Form Quality of Life. Higher scores are better (higher quality of life) and lower scores are worse (poorer quality of life). score range 0-100.
Time Frame: 12 months
Population: At 12 months in the hypnotherapy group: 4 had withdrawn, 1 missing diary. In the medication group, 7 had withdrawn.
Measure: Least Squares Mean (95% Confidence Interval); unit: sub-scale scores
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 69 | 71
sub-scale scores | 75.71 [68.07 to 83.35] | 81.57 [74.91 to 88.23]

10. Secondary Outcome: Voids on Bladder Diary
Description: Total Number of voids on 3-day bladder diary.
Time Frame: 2 months
Population: At 2 months in the hypnotherapy group of the 74 randomized, 3 had withdrawn and 1 was lost. In the medication group, of 78 randomized: 4 had withdrawn and 2 were missing diaries.
Measure: Mean (95% Confidence Interval); unit: counts
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 70 | 72
counts | 26.4 [24.29 to 31.08] | 25.35 [23.59 to 27.12]

11. Secondary Outcome: Voids on Bladder Diary
Description: number of voids on 3-day bladder diary
Time Frame: 6 months
Population: Of the 74 women randomized to hypnotherapy, at 6 months: 4 had withdrawn and 2 were lost and 1 was missing diary information. Of the 78 women randomized to medications, 6 had withdrawn and 1 was lost.
Measure: Mean (95% Confidence Interval); unit: counts
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 67 | 71
counts | 25.58 [23.48 to 27.68] | 24.28 [22.69 to 25.87]

12. Secondary Outcome: Voids on Bladder Diary
Description: number of voids on 3-day bladder diary
Time Frame: 12 months
Population: At 12 months, of the 74 randomized to hypnotherapy: 4 had withdrawn and 1 was missing diary information. Of the 78 women randomized to medications, 7 had withdrawn.
Measure: Mean (95% Confidence Interval); unit: counts
Arm/Group | Hypnotherapy | Anticholinergic Medications
Number analyzed (Participants) | 69 | 71
counts | 25.74 [23.69 to 27.79] | 25.37 [23.71 to 27.02]

ADVERSE EVENTS:
Time Frame: 1 year; from study randomization to study completion
Description: Adverse event collection occurred at all follow-up and by spontaneous participant report
Arm/Group | Hypnotherapy | Anticholinergic Medications
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/70 | 3/72
Other Adverse Events (participants affected / at risk) | 12/70 | 27/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypnotherapy (N=70) | Anticholinergic Medications (N=72)
1 inpatient hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0) — admitted with worsening hyperparathyroidism; a pre-existing condition
1 inpatient hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — fell off horse when horse stepped into a hole and incurred trauma to leg.
1 inpatient hospitalization for observation (Cardiac disorders) | 0 (0) | 1 (1) — pt had abnormal cardiac stress test with pre-existing cardiac disease. Patient's cardiac work up in the hospital was negative
1 in-patient hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — pt had pre-existing chronic back pain. Hospitalized for possible disc disease. Recovered and returned to usual activities with continued follow-up with orthopedic physician.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypnotherapy (N=70) | Anticholinergic Medications (N=72)
Falls (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) — Fell on floor
urinary tract infection (Infections and infestations) | 5 (5) | 6 (6) — treated for urinary tract infection
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) — complaint of back pain
expected adverse events pharmacotherapy (General disorders) | 1 (1) | 12 (12) — dry eyes, dry mouth, constipation, dyspepsia These expected events were not gathered separately and are therefore are listed together

LIMITATIONS AND CAVEATS:
Women willing to participate x1 yr in RCT may not represent the general population. Population limited to 1 U.S. southwestern institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT01829425/Prot_SAP_000.pdf